CLINICAL TRIAL: NCT02356315
Title: Investigating Pain Processing in the Brain, Brainstem, and Spinal Cord With fMRI
Brief Title: Brain, Brainstem, and Spinal Cord fMRI
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Todd Parrish, Professor, Department of Radiology, Northwestern University
Other Study IDs: STU00067625; 5F32AT007800-03 (NIH)
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Neck Pain; Chronic Pain
Keywords: Brain; Brain Stem; Spinal Cord; Neurophysiology; Magnetic Resonance Imaging
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy subjects: Functional magnetic resonance imaging of healthy subjects
  Interventions: Other: Functional Magnetic Resonance Imaging
- Chronic neck pain patients: Functional magnetic resonance imaging of chronic neck pain patients
  Interventions: Other: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging — Functional magnetic resonance imaging will be performed to measure brain, brainstem, and spinal cord activity.

SUMMARY:
New advances in medical imaging have allowed for the measurement of brain activity related to chronic pain. In addition to the brain, the investigators aim to use functional magnetic resonance imaging to investigate pain processing in the brainstem and spinal cord in healthy subjects and chronic neck pain patients. The information gained from this study will increase the investigators understanding of how chronic pain is encoded in the nervous system and assist in developing more effective treatment strategies.

DETAILED DESCRIPTION:
The experimental design is an observational (non-interventional) cross-sectional clinical study. The principal goal of the proposed research is to utilize functional magnetic resonance imaging to further investigate and characterize pain-related neural activity at the level of the brain, brainstem, and spinal cord in healthy subjects and chronic neck pain patients. Healthy subjects and chronic neck pain patients will be recruited and participate in a single session of data collection. For both the healthy and chronic neck pain groups, painful thermal stimuli will be applied over the skin of the upper extremity while whole brain, brainstem, and cervical spinal cord functional images are acquired (on separate scans). For the chronic neck pain group, additional scans (brain, brainstem, and cervical spinal cord) will be acquired while the subjects rate their spontaneous chronic neck pain.

ELIGIBILITY:
Healthy subjects must meet all of the following inclusion criteria to participate in this study:

1. Age between 21 and 60 years old
2. Right-handed; not currently experiencing significant pain
3. No history of a chronic pain syndrome such as fibromyalgia, complex regional pain syndrome, chronic low back pain, etc.

Chronic neck pain patients must meet all of the following inclusion criteria to participate in this study:

1. Age between 21 and 60 years old
2. Right handed; neck pain > 3 months duration; moderate neck pain score > 30 on VAS (0-100) 3) No history of a chronic pain syndrome (fibromyalgia, complex regional pain syndrome, chronic low back pain, etc.) other than chronic neck pain and its associated symptoms.

Participants meeting any of the following exclusion criteria at baseline will be excluded from study participation:

1. Non-English speaking
2. Signs of upper extremity sensation loss; history of significant cerebrovascular disease including (but not limited to) epilepsy, stroke, tumor, multiple sclerosis, meningitis
3. History of major head trauma with sustained loss of consciousness; history of neurosurgery, ENT surgery, spine surgery, or cardiac surgery
4. History of cardiac pacemaker or neurostimulator implantation
5. History of significant medical illness including cardiovascular disease, uncontrolled diabetes, uncontrolled hypertension, cancer, chronic obstructive pulmonary disease, severe asthma requiring hospitalization for treatment, renal insufficiency requiring dialysis, etc.
6. History of alcoholism or consistent drug use; current infection or fever; pregnancy (or possible pregnancy)
7. History of metal working or injury with shrapnel or metal slivers
8. Claustrophobia
9. Piercings that are unable to be removed and tattoos older than 30 years

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects and chronic neck pain patients recruited from the community
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging | 1.5-2.25 hours
  Use functional magnetic resonance imaging to characterize brain, brainstem, and spinal cord pain processing in healthy subjects (thermal pain) and chronic neck pain patients (thermal pain and spontaneous clinical pain).

CONTACTS AND LOCATIONS:
Overall Officials: Todd Parrish, PhD, Principal Investigator — Northwestern University
Locations (1):
- Center for Translational Imaging, Northwestern University, Chicago, Illinois, United States